CLINICAL TRIAL: NCT04260035
Title: The Effects of a Long-lasting Infusion of Vasoactive Intestinal Peptide (VIP) on Headache, Cranial Hemodynamic and Autonomic Symptoms in Episodic Migraine Patients Without Aura
Brief Title: The Effects of a Long-lasting Infusion of Vasoactive Intestinal Peptide (VIP) in Episodic Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Lanfranco Pellesi, Principal Investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-19075630
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Migraine; Pain; Neurologic Manifestations; Signs and Symptoms; Brain Diseases; Central Nervous System Diseases
MeSH Terms: conditions — Migraine Disorders; Pain; Neurologic Manifestations; Signs and Symptoms; Brain Diseases; Central Nervous System Diseases | interventions — Vasoactive Intestinal Peptide; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vasoactive Intestinal Polypeptide (VIP) (Active Comparator): Intravenous infusion of 8 pmol/Kg/min of Vasoactive Intestinal Polypeptide (VIP).
  The infusion is administered at constant speed by an automatic pump, lasting 120 minutes.
  Interventions: Drug: Vasoactive Intestinal Polypeptide (VIP)
- Sterile, isotonic, non-active saline (Placebo) (Placebo Comparator): Intravenous infusion of sterile, isotonic, non-active saline 9 mg/ml (placebo). The infusion is administered at constant speed by an automatic pump, lasting 120 minutes.
  Interventions: Drug: Sterile saline

INTERVENTIONS:
Drug: Vasoactive Intestinal Polypeptide (VIP) — 20 episodic migraine patients without aura of both genders are randomized to receive a 2-hour infusion of VIP and/or sterile saline on two days, with at least one week in between.
  Other Names: Vasoactive Intestinal Peptide (VIP)
  Arms: Vasoactive Intestinal Polypeptide (VIP)
Drug: Sterile saline — 20 episodic migraine patients without aura of both genders are randomized to receive a 2-hour infusion of VIP and/or sterile saline on two days, with at least one week in between.
  Other Names: Isotonic saline; 0.9% saline
  Arms: Sterile, isotonic, non-active saline (Placebo)

SUMMARY:
Vasoactive intestinal peptide (VIP) is a peptide of 28 amino acid residues that belongs to the glucagon/secretin superfamily of peptides. Along with other neuropeptides, such as calcitonin gene-related peptide (CGRP) and pituitary adenylate cyclase-activating polypeptide (PACAP), it is released from the trigeminal afferents and exerts a strong vasodilating activity on the cranial vasculature. Especially, it shares 70% structure with PACAP and acts on the same receptors. But, unlike it, VIP cannot induce a long-lasting vasodilation and has a modest capability to induce migraine attacks. Whether it may induce migraine-like attacks in migraine patients, as a twenty-minute infusion of PACAP, is unknown.

DETAILED DESCRIPTION:
The vasoactive intestinal polypeptide (VIP) is a peptide of 28 amino acid residues that belongs to the glucagon/secretin superfamily of peptides. It is distributed in different regions of the nervous system, including several autonomic ganglia and the brain. Once released from neurons, it acts on the vasoactive intestinal peptide receptor 1 (VPAC1), the vasoactive intestinal peptide receptor 2 (VPAC2) and the pituitary adenylate cyclase-activating polypeptide type I receptor (PAC1). All three belong to a family of G-protein coupled receptors, sharing the activation of adenylate cyclase and the increase in intracellular cyclic adenosine monophosphate (cAMP). The three receptors are involved in many physiological functions, among them the vasodilating and parasympathetic responses. VPAC1 and VPAC2 are expressed in dura mater vessels and are primarily responsible for the relaxation of arteries. PAC1 is located in the trigemino-autonomic system, but not in blood vessels. VIP shares the binding to the three aforementioned receptors with other peptides, including the pituitary adenylate cyclase-activating polypeptide-38 (PACAP38), and the pituitary adenylate cyclase-activating polypeptide-27 (PACAP27).

20-minute infusion of VIP and PACAPs in patients with migraine dilated cranial arteries. However, only PACAP27 and PACAP38 induced a sustained cranial vasodilation, and migraine like-attacks. VIP-induced cranial vasodilation was of short duration, and patients did not report migraine-like attacks. The discrepancy was ascribed to the preferential activation of the PAC1 receptor by PACAPs, but a monoclonal antibody against PAC1 receptor recently failed in migraine prevention. Currently, it is unknown whether the prolonged cranial vasodilation related with the appearance of migraine-like attacks. More recently, a two-hour infusion of VIP promoted a long-lasting cranial vasodilation and delayed headache in healthy volunteers, resembling the effect of PACAP27 and PACAP38, two closely related peptides causing migraine. Whether a long-lasting infusion of VIP may induce a sustained cranial vasodilation and migraine-like attacks in migraine patients, as a twenty-minute infusion of PACAP27 and PACAP38, is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine without aura as according to the International Classification
* Frequency of migraine attacks between one and six attacks within 8 weeks
* Weight: 50-90 kg
* Fertile women should use contraception. Fertile women do not include hysterectomies women or women who are postmenopausal for at least 2 years. Contraception includes either IUD, birth control pills, surgical sterilization of the woman or depot progesterone

Exclusion Criteria:

* Any other type of headache (including > 2 days of tension-type headache per month)
* Headache less than 48 hours before the start of the experiment
* Daily intake of any medicine other than oral contraception
* Pregnant or breastfeeding women
* Clinical signs of Hypertension (systolic blood pressure > 150 mmHg and / or diastolic blood pressure > 100 mmHg) and/or Hypotension (systolic blood pressure < 90 mm Hg and / or diastolic blood pressure < 50 mmHg)
* Cardiovascular disease of all kinds, including cerebrovascular disease
* Anamnestic or clinical signs of mental illness, abuse or smoking

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of migraine-like attacks | Before (-10 minutes) and after the drug administration (+12 hours)
  Migraine-like attack fulfilling either (i) or (ii):
  (i) Headache fulfilling criteria C and D for migraine without aura according to the International Classification od Headache Disorders: C. Headache has at least two of the following four characteristics: unilateral location; pulsating quality; moderate or severe pain intensity (moderate pain intensity is considered 5 or 4 on verbal rating scale); aggravation by cough (hospitalization phase) or causing avoidance of routine physical activity (out-hospital phase); D. During headache at least one of the following: nausea and/or vomiting; photophobia and phonophobia; (ii) Headache described as mimicking the patient's usual migraine attack and treated with acute migraine medication (rescue medication).

SECONDARY OUTCOMES:
Change in cranial hemodynamic | Before (-10 minutes) and after the drug administration (+3 hours)
  Change on diameter (mm) of superficial temporal artery (STA)
Occurrence of headache and change of headache intensity scores | Before (-10 minutes) and after the drug administration (+12 hours)
  Headache intensity scores are measured by a numerical rating scale (NRS). It is a verbally declared scale from 0 to 10, where 0 is no headache; 1 is a very mild headache, including a feeling of pressing or throbbing; 5 is a moderate headache; 10 is the worst imaginable headache.
Change in Mean Arterial Pressure | Before (-10 minutes) and after the drug administration (+3 hours and 20 minutes)
  Blood pressure was measured using an auto-inflatable cuff (Protocol, Oregon, USA). Blood pressure was registered as mean arterial pressure (MAP), equal to diastolic blood pressure + 1/3 (systolic blood pressure - diastolic blood pressure).
Change in Heart Rate | Before (-10 minutes) and after the drug administration (+3 hours and 20 minutes)
  Heart rate was measured using an auto-inflatable cuff (Protocol, Oregon, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, PhD, Study Director — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pellesi L, Al-Karagholi MA, De Icco R, Chaudhry BA, Lopez CL, Snellman J, Hannibal J, Amin FM, Ashina M. Plasma Levels of CGRP During a 2-h Infusion of VIP in Healthy Volunteers and Patients With Migraine: An Exploratory Study. Front Neurol. 2022 Apr 1;13:871176. doi: 10.3389/fneur.2022.871176. eCollection 2022. PMID 35432170
- [Derived] Pellesi L, Al-Karagholi MA, De Icco R, Coskun H, Elbahi FA, Lopez-Lopez C, Snellman J, Hannibal J, Amin FM, Ashina M. Effect of Vasoactive Intestinal Polypeptide on Development of Migraine Headaches: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2118543. doi: 10.1001/jamanetworkopen.2021.18543. PMID 34357396